CLINICAL TRIAL: NCT00838838
Title: Nebido® Therapy in Hypogonadal Male Patients With Osteoporosis Associated With Paraplegia Compared With Conventional Osteoporosis - Prophylaxis / Therapy in Hypogonadal and Eugonadal Patients With Osteoporosis Associated With Paraplegia
Brief Title: Efficacy of Nebido on Bone Mineral Density (BMD) in Hypogonadal Paraplegic Patients With Confirmed Osteoporosis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 13900; NE0501
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Hypogonadism; Paraplegia; Bone Density; Osteoporosis
Keywords: Testosterone replacement therapy; Hypogonadism; Osteoporosis; Immobilisation; Paraplegia; Testosterone
MeSH Terms: conditions — Hypogonadism; Paraplegia; Osteoporosis | interventions — Testosterone Propionate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Testosterone Undeconate (Nebido-R, BAY86-5037)

INTERVENTIONS:
Drug: Testosterone Undeconate (Nebido-R, BAY86-5037) — Male patients > 18yrs in medical practices fulfilling all criteria for documentation.

SUMMARY:
Both conditions hypogonadism and immobilisation (paraplegia) may contribute or lead to decreased bone mineral density resp osteoporosis. In this study bone mineral density is assessed in hypogonadal paraplegic patients, who are on standard prophylactic therapy for osteoporosis and and on a standard physiotherapy exercise program one group receiving Nebido for testosterone replacement (TRT). The additional effect of TRT on bone mineral density / osteoporosis is assessed (CT scan lumbar spine).

ELIGIBILITY:
Inclusion Criteria:

* Male patients > 18yrs
* Osteoporosis prophylaxis/therapy with

  * vitamin D 800 - 1200 mg per day,
  * calcium 800 - 1000 mg per day,
  * Fosamax 70 once a week.
* Standardised physiotherapy exercise programme.
* No proliferative bone disease.
* No history of calcium oxalate stones.
* No use of aromatase inhibitors.
* No use of 5-alpha reductase inhibitors.

Nebido group:

* No contraindications to use of Nebido (known prostate or breast carcinoma or suspicion thereof, no past or present history of liver tumours);
* No known hypersensitivity to testosterone or excipients of Nebido

Exclusion Criteria:

* Androgen dependent carcinoma of the prostate or male mammary gland, past or present history of liver tumours, hypersensitivity towards the active pharmaceutical ingredient or other ingredients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients > 18yrs in medical practices fulfilling all criteria for documentation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (CT lumbar spine) | 12 weeks after 4th injection

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany